CLINICAL TRIAL: NCT01522729
Title: Impact of Somatosensory Feedback on Peripheral Muscle Fatigue and Exercise Tolerance in Patients With COPD
Brief Title: Impact of Muscle Afferent Feedback During Exercise in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Philippe Gagnon, PhD Candidate, PhD Candidate, Laval University
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: SPINAL-20520
Record Dates: First submitted 2012-01-20; First posted 2012-02-01 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic pulmonary obstructive disease; Muscle dysfunction; Exercise intolerance; Muscle afferents; Ventilation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Aspiration | interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fentanyl (Experimental)
  Interventions: Drug: Fentanyl
- Placebo (Experimental)
  Interventions: Drug: Placebo comparator

INTERVENTIONS:
Drug: Fentanyl — Single-dose of intrathecal fentanyl [25ug] Duration of fentanyl : 3.5 hours
  Arms: Fentanyl
Drug: Placebo comparator — placebo [NaCl]
  Arms: Placebo

SUMMARY:
Recently, direct evidences point to the contributing role of peripheral muscle fatigue in exercise tolerance among patients with COPD. However, the physiological mechanisms by which peripheral muscle fatigue impairs exercise tolerance are still unknown, as factors regulating peripheral muscle fatigue in COPD may be complex. One possible link between limb muscle fatigue and exercise intolerance could be enhanced afferent signals from the active limb muscles to the central command, thereby limiting central motor output and eventually leading to exercise termination.

A direct method to investigate the regulation of peripheral muscle fatigue during exercise in patients with COPD is the blockade of peripheral neural afferents via lumbar anesthesia. Consequently, investigating the interplay between the peripheral muscular component and the central motor command during self-paced exercise could shed light on the regulation of peripheral muscle fatigue in COPD and its implication in exercise intolerance.

DETAILED DESCRIPTION:
The aim of the study is to characterize the role of peripheral muscle afferents on the development of muscle fatigue, cardiorespiratory response and exercise tolerance to constant-workrate endurance cycling exercise in patients with COPD.

In a double-blind randomized design, patients with GOLD stage II-III COPD will be recruited and will complete a constant-workrate cycling test following either the injection of a placebo [NaCl, interspinous L2-L3] or an opioid [Fentanyl 25 µg, intrathecal L2-L3] inhibiting central feedback of peripheral muscles sensory afferents. Quadriceps force (TwQ) will be measured by magnetic stimulation of the femoral nerve and central chemoreceptors response will be assessed by CO2 rebreathing, both performed before and after the injection. Finally, TwQ will also be measured after the endurance cycling test to assess the magnitude of quadriceps fatigue induced by symptom-limited exercise.

ELIGIBILITY:
Inclusion Criteria:

* Smoking history > 15 pack-years
* COPD GOLD II-III (30 % predicted < FEV1 < 80 % predicted; FEV1/FVC < 0.70)

Exclusion Criteria:

* Unstable condition
* Recent exacerbation (<3 months)
* Recent cancer (<3 months)
* Myopathy, neuromuscular disease
* Unstable cardiac disease
* Hepatic, kidney, intestinal disease
* BMI > 35
* PaCO2 > 45 mmHg
* PaO2 < 60 mmHg

Ages: 55 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Endurance time | 60-min post-anesthesia - From the start to the end of the constant-workload cycling test (limited by symptoms of the patients)
  Exercise tolerance is referred as the endurance time (sec) during constant-workrate cycling test at 80 % of the predetermined maximal workload in every conditions (placebo and fentanyl)

SECONDARY OUTCOMES:
Ventilatory response | 60-min post-anesthesia-From the start to the end of the constant-workload cycling test (limited by symptoms of the patients)
  The ventilatory response (Ventilation, L/min) will be monitored continuously during the cycling test and will be compared between the two conditions (placebo vs. fentanyl)
Quadriceps muscle fatigue | 15-min after the end of constant-workload cycling test
  The quadriceps muscle fatigue will be monitored before and after the cycling test to quantify the extent of muscle fatigue produced by the cycling test. This will be done by magnetic stimulation of the femoral nerve and maximal voluntary contraction. Also, non-invasive surface electromyography (EMG) of the quadriceps will help to better characterize muscle fatigue.
Dynamic hyperinflation | 60-min post-anesthesia-From the start to the end of the constant-workload cycling test (limited by symptoms of the patients) - Every 2-min during exercise
  Dynamic hyperinflation will be monitored periodically every 2-min during the cycling test by manoeuvres of inspiratory capacity and will be compared between the two conditions (placebo vs. fentanyl)
Effort perception | 60-min post-anesthesia-From the start to the end of the constant-workload cycling test (limited by symptoms of the patients) - Every 2-min during exercise
  Leg fatigue and dyspnea perception (Borg scale scores) will be monitored periodically every 2-min during the cycling test and will be compared between the two conditions (placebo vs. fentanyl)

CONTACTS AND LOCATIONS:
Overall Officials: François Maltais, MD, Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Locations (1):
- Institut universitaire de cardiologie et de pneumologie de Québec - Université Laval, Québec, Quebec, Canada

REFERENCES:
- [Derived] Gagnon P, Bussieres JS, Ribeiro F, Gagnon SL, Saey D, Gagne N, Provencher S, Maltais F. Influences of spinal anesthesia on exercise tolerance in patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2012 Oct 1;186(7):606-15. doi: 10.1164/rccm.201203-0404OC. Epub 2012 Jul 19. PMID 22822019